CLINICAL TRIAL: NCT03162809
Title: Venopuncture-Free Monitoring During IVF: Are More Frequent Sequential Salivary Hormone Measurements More Informative Than Daily Serum Monitoring of IVF Patients?
Brief Title: Needle-Free Monitoring for IVF Patient Cycles
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Boston IVF (Other)
Responsible Party: Sponsor
Other Study IDs: SAL201702
Record Dates: First submitted 2017-04-11; First posted 2017-05-22 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Infertility
Keywords: infertility; in vitro fertilization; Estradiol; Progesterone
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Salivary diagnostic testing is emerging as a less invasive, inexpensive alternative to serum analyte measurements with proven diagnostic accuracy in clinical settings. This study aims to continue analyzing aspects of the performance of salivary hormone competitive immunoassays for monitoring patient's reproductive hormone profiles in the reproductive cycle. Hormone levels will be monitored during treatment cycles for infertility.

DETAILED DESCRIPTION:
This study will be a prospective study to measure salivary and serum estrogen and progesterone levels in subject's voluntarily undergoing monitored infertility treatment cycles including controlled ovarian stimulation (COS) with oral agents or gonadotropins and controlled ovarian hyperstimulation (COH) for in vitro fertilization (IVF). Ultimately, the potential applicability and reliability of salivary steroid monitoring in IVF cycles will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of infertility.
* Cycle start age of 25 -43 years.
* Undergoing controlled ovarian stimulation for IVF.
* All monitoring scheduled at the participating IVF facility.

Exclusion Criteria:

-Prior cancelled cycle due to hyperstimulation.

Ages: 25 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients undergoing In Vitro Fertilization (IVF) at a participating infertility center
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-05-09 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Measurement of multiple Progesterone levels as an aid during an IVF cycle | 1 month
  To determine if collecting multiple salivary Progesterone levels versus a single serum hormone sample could assist in predicting the administration of Human Chorionic Gonadotropin (HCG) during an IVF cycle.

SECONDARY OUTCOMES:
Measurement of salivary Estradiol level as an aid during fertility treatment | 1 month
  Comparison of salivary reproductive hormone values versus serum collection to see if there is a correlation between the two methods of collection.
Measurement of salivary Progesterone level as an aid during fertility treatment | 1 month
  Comparison of salivary reproductive hormone values versus serum collection to see if there is a correlation between the two methods of collection.

CONTACTS AND LOCATIONS:
Overall Officials: Denny Sakkas, PhD, Principal Investigator — Boston IVF
Locations (1):
- Boston IVF, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No